CLINICAL TRIAL: NCT05688813
Title: Comparison of Caudal Block and Sacral Erector Spinae Block for Postoperative Analgesia in Circumcision in Pediatric Patients: A Double-blind, Randomized Controlled Trial
Brief Title: Comparison of Caudal Block and Sacral Erector Spinae Block for Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Volkan Ozen, Associate Professor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021.51
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Pain; Children, Only
Keywords: Ultrasound; Pain; Sacral erector spinae block; Caudal block
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: A nurse was blinded to collect the pain score. An anesthesiologist was blinded to data collection about the analgesic requirements and postoperative complications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal block group (Experimental): An echogenic block needle (22 Gauge 50 mm) was then advanced into the sacral canal through the sacrococcygeal membrane while a longitudinal position was used, continuing with the in-plane technique. After ensuring that there is no blood or cerebrospinal fluid with aspiration, 0.5 ml/kg 0.25% bupivacaine was administered while observing caudal epidural space dilation or turbulent flow with Doppler.
  Interventions: Procedure: Regional anesthesia intervention
- Sacral erector spinae block (Experimental): Following antiseptic preparation of block site linear ultrasound probe was placed longitudinally to midline just above the sacrum. After the median sacral crests and erector spinae were identified, a 22G, 50 mm block needle was advanced from the cranial to the caudal direction until it touched the top of the 4th median sacral crest with the in-plane technique. After hydrodissection was achieved with 1 ml of saline, 0.5 ml/kg of 0.25% bupivacaine was administered after negative aspiration.
  Interventions: Procedure: Regional anesthesia intervention

INTERVENTIONS:
Procedure: Regional anesthesia intervention — Ultrasound-guided caudal and sacral erector spinae blocks were administered

SUMMARY:
Caudal block (CB) has been the method used for years to achieve adequate postoperative analgesia in pediatric patients, which is one of the main responsibilities of an anesthetist. CB, which has been proven to provide effective analgesia for many different indications, is the most commonly performed neuraxial block technique for postoperative pain control in urogenital surgeries. However, in the following years, truncal nerve blocks are recommended for postoperative analgesia by the literature both for more effective analgesia and for preventing complications of CB that may prevent early mobilization and prolong hospital discharge

DETAILED DESCRIPTION:
Circumcision, which is widely performed in male children for cultural and religious reasons in our country, is one of the daily urological surgical procedures with painful postoperative period. However, in the following years, truncal nerve blocks are recommended for postoperative analgesia by the literature both for more effective analgesia and for preventing complications of CB that may prevent early mobilization and prolong hospital discharge. Based on this knowledge, in order to provide postoperative analgesia in urogenital surgeries in male children sacral ESP (SESP) block can be used as an alternative to CB due to its undesirable effects

ELIGIBILITY:
Inclusion Criteria:

* 1-7 years of age
* ASA (American Society of Anesthesiologists) I-II group
* Scheduled for circumcision
* Able to communicate in Turkish
* Willing to participate to the study (parents and children)

Exclusion Criteria:

* Less than 1 or more than 7 years of age
* A neurological deficit, bleeding diathesis, or a history of local anesthetic allergy; an infection or redness in the injection area, congenital lumbar anomaly, liver and/or kidney disorder, a psychiatric disorder, mental retardation, or communication problems detected during examination
* Unwilling to to participate to the study ((parents or children)

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Analgesic efficiency | Up to 24 hours
  The analgesic efficacy was evaluated based on postoperative pain scores via Face, Legs, Activity, Cry, Consolability (FLACC) scale. The lowest scale score is 0 points and the highest 10 points

SECONDARY OUTCOMES:
Time of Postoperative analgesic requirement | Up to 24 hours
  It was assessed five times after the operation with Face, Legs, Activity, Cry, Consolability (FLACC) scale. The lowest scale score is 0 points and the highest 10 points. Significant pain behavior for the scale has been identified as 4 points or more. Following transfer from the recovery unit to the ward, the 30 minutes, 1st, 2nd, 4th, and 6th hour pain levels were evaluated by the ward nurse. Paracetamol was administered IV at a dose of 10 mg/kg if the scale score was 4 or higher
Rate of Postoperative complications | Up to 6 hours
  The presence of urinary retention, motor block, and ecchymosis or hematoma at the injection site was evaluated in the postoperative period by the anesthesiologist who was blind to the study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aksu C, Sen MC, Akay MA, Baydemir C, Gurkan Y. Erector Spinae Plane Block vs Quadratus Lumborum Block for pediatric lower abdominal surgery: A double blinded, prospective, and randomized trial. J Clin Anesth. 2019 Nov;57:24-28. doi: 10.1016/j.jclinane.2019.03.006. Epub 2019 Mar 6. PMID 30851499
- [Background] Ozen V, Yigit D. A Comparison of the Postoperative Analgesic Effectiveness of Ultrasound-Guided Dorsal Penile Nerve Block and Ultrasound-Guided Pudendal Nerve Block in Circumcision. Urol Int. 2020;104(11-12):871-877. doi: 10.1159/000509173. Epub 2020 Aug 13. PMID 32791500
- [Background] Desai N, Chan E, El-Boghdadly K, Albrecht E. Caudal analgesia versus abdominal wall blocks for pediatric genitourinary surgery: systematic review and meta-analysis. Reg Anesth Pain Med. 2020 Nov;45(11):924-933. doi: 10.1136/rapm-2020-101726. Epub 2020 Sep 14. PMID 32928996